CLINICAL TRIAL: NCT00852904
Title: Vanguard Phase of the National Children s Study
Brief Title: National Children s Health Study
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909083; 09-CH-N083
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Infant; Child Development; Biological Samples
Keywords: Childhood Growth and Development; Genetics; Children; Environment; Longitudinal Study; National Children's Study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- NCS Vanguard cohort: Women of child bearing potential, children born to women enrolled in the study, the children s biological and/or social fathers, and primary caregivers (if other than parent)

SUMMARY:
Patterns of illness among children in the United States and other industrially developed nations have changed substantially during the past 100 years. Before and during the first half of the previous century, infectious diseases were the primary threat to children s health. In contrast, the major illnesses and disorders that impair health, growth, and development today are chronic conditions stemming from the complex interaction of environmental exposures and inherent genetic factors. The Children s Health Act of 2000 directed the National Institute of Child Health and Development to conduct a national longitudinal study of environmental influences on children s health in the United States. The act specified that the study extend from the prenatal period to adulthood and investigate the short-term and long-term influences of physical, chemical, biological, and psychosocial environmental exposures on children s health and development, including behavioral, emotional, and educational outcomes in addition to physical health. The National Children s Study (NCS) is an observational longitudinal study that will enroll and follow a nationally representative sample of approximately 100,000 U.S.-born children from before birth through their 21st birthday. The study will screen all households within selected areas of 105 locations (primarily counties).

The major types of analysis of NCS data will include longitudinal exposure-outcome analysis, identification of causal pathways, analysis of neighborhood effects, evaluation of temporal effects within longitudinal data analysis of data from case-control data, and analysis of genomic data.

Women in their first trimester of pregnancy will be invited to participate in the pre-pregnancy portion of the NCS. Women who are not pregnant but have a high probability of becoming pregnant will be asked to participate in the early pregnancy portion of the NCS. All other eligible women will be asked if the study can contact them periodically to assess their pregnancy status. They also will be asked to contact the NCS should they become pregnant. Women identified as pregnant within 4 years after initial screening will be invited to enroll in the NCS.

The following information will be gathered:

Mother s data and information

* Questionnaire data interviewed and self-administered (e.g., demographics; current pregnancy history; reproductive history; medical conditions; health behaviors; doctor visits; medicines and supplements; housing characteristics; pesticides, product use; occupation, hobbies; depression, stress; social support; diet; time and activity)
* Physical measures and clinical data (e.g., blood pressure, sonograms, height, weight, body measurements)
* Biologic specimens (e.g., blood, urine, hair, saliva)
* Environmental samples during home visits (e.g., dust, air, water)
* Medical record abstraction

Infant s data and information at birth

* Cord blood and tissue samples of the placenta and umbilical cord
* Standardized neurobehavioral exam
* Physical measures and clinical data (e.g., length; weight; circumferences of head, arm, abdomen, thigh)
* Meconium samples
* Medical diagnoses and treatment by report
* Selected Medical record abstraction

DETAILED DESCRIPTION:
The National Children s Study (NCS) is a planned, observational, and longitudinal study that will enroll and follow a national sample of approximately 100,000 children born in the United States (US) to participating women from before birth through the child s 21st birthday. The goal of the NCS is to provide information that will ultimately lead to improvements in the health, development, and well-being of children. The primary aim of the NCS is to investigate the separate and combined effects of environmental exposures (chemical, biological, physical, and psychosocial) as well as gene-environment interactions on pregnancy outcomes, child health and development, and precursors of adult disease. In-person contacts with the NCS participants include visits during pregnancy, after delivery, and throughout infancy and childhood at the participant s home and sometimes in a clinical setting. The collection of biospecimens, environmental samples, and physical measures is involved in addition to the examination of the infant and periodic contacts with the family. In addition, interim phone interviews regularly occur with in-person contacts. The NCS consists of the NCS Vanguard Study with any sub-studies and the NCS Main Study with any sub-studies. The Vanguard Study is the precursor to the Main Study.

The NCS Vanguard Study is designed and implemented to determine the feasibility, acceptability and cost of the elements that will form the Main Study. The Vanguard Study enrolls participants at forty Study locations and will have a planned duration of 21 years following completion of enrollment. The Vanguard Study will precede the Main Study on an ongoing basis to pilot all aspects of the Main Study. The specific objectives of the Vanguard Study are:

1. Evaluation of recruitment, enrollment and retention strategies
2. Evaluation of study logistics and operations including sites and mechanisms of data acquisition, collection, transport and storage of environmental and biological samples, and design and performance of information systems
3. Evaluation of study visit assessments for feasibility, acceptability, reliability, reproducibility, cost, value, stability, and redundancy with other assessments

Families who participate in the NCS will come from forty Study locations across the US. Study visit assessments are the tests, environmental samples, biospecimens, questionnaires and other forms of data acquisition that are scheduled at the study visits. The evaluation of the Vanguard Study will be based on a series of targeted and specific statistical techniques and tests selected for each evaluation. Multiple performance measures will be used to inform the scope, design, visit structure and schedule, mechanisms and procedures, and analysis plan for the Main Study.

ELIGIBILITY:
* IINCLUSION CRITERIA:
* Women age 18-49 years of age at the time of enumeration who medically could be pregnant
* Pregnant women at or above the local age of majority
* During the Initial Vanguard Study recruitment period only: pregnant women aged younger than 18, residing in a selected NCS geographic segment at the time of enrollment, who are considered to be emancipated minors per the laws of their jurisdiction or minor pregnant women who obtain parental consent for participation
* Children born to enrolled women
* Biological and social fathers as identified by enrolled women
* Adult guardians who have legal responsibility to authorize needed care for enrolled children
* Adults who are primary caregivers of enrolled children

EXCLUSION CRITERIA:

* Women self-reported to be infertile
* Adults who are unable to understand what is involved in NCS participation and grant informed consent
* Prisoners as defined in 45 CFR 46.303[c]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women of child bearing potential, their children, the children's biological and/or ocial fathers, and primary caregivers (if other than parent)
Sampling Method: Non-Probability Sample
Enrollment: 9942 (Actual)
Dates: Start 2009-02-25 (Actual); Primary Completion 2014-12-12 (Actual); Study Completion 2020-05-29 (Actual)

PRIMARY OUTCOMES:
Assess feasibility, acceptability and cost of: Recruitment, accrual, enrollment and retention strategies; Study logistics and operations; Study visit assessments including newly developed assessmentsfor reliability, reproducibility and stabil... | During and after pregnancy, throughout infancy and childhood until age 21
  Feasibility, acceptability and cost of the elements that will form the Main Study

SECONDARY OUTCOMES:
Evaluation of recruitment, enrollment and retention strategies | Ongoing
  Recruitment, enrollment and retention

CONTACTS AND LOCATIONS:
Overall Officials: Jack Moye, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (4):
- United States (4):
  - Northwestern University, Chicago, Illinois
  - NORC at the Univ. of Chicago, Chicago, Illinois
  - National Institute of Child Health and Human Development (NICHD), 9000 Rockville, Bethesda, Maryland
  - Westat, Inc., Rockville, Maryland

REFERENCES:
- [Background] Hudak ML, Park CH, Annett RD, Hale DE, McGovern PM, McLaughlin TJ, Dole N, Kaar JL, Balsam MJ. The National Children's Study: An Introduction and Historical Overview. Pediatrics. 2016 Jun;137 Suppl 4(Suppl 4):S213-8. doi: 10.1542/peds.2015-4410B. PMID 27251867
- [Background] Li Q, Kappil MA, Li A, Dassanayake PS, Darrah TH, Friedman AE, Friedman M, Lambertini L, Landrigan P, Stodgell CJ, Xia Y, Nanes JA, Aagaard KM, Schadt EE, Murray JC, Clark EB, Dole N, Culhane J, Swanson J, Varner M, Moye J, Kasten C, Miller RK, Chen J. Exploring the associations between microRNA expression profiles and environmental pollutants in human placenta from the National Children's Study (NCS). Epigenetics. 2015;10(9):793-802. doi: 10.1080/15592294.2015.1066960. Epub 2015 Aug 7. PMID 26252056
- [Background] Park CH, Winglee M, Kwan J, Andrews L, Hudak ML. Comparison of Recruitment Strategy Outcomes in the National Children's Study. Pediatrics. 2017 Aug;140(2):e20162822. doi: 10.1542/peds.2016-2822. PMID 28724571
- [Derived] Gilbertson PK, Forrester S, Andrews L, McCann K, Rogers L, Park C, Moye J. The National Children's Study Archive Model: A 3-Tier Framework for Dissemination of Data and Specimens for General Use and Secondary Analysis. Front Public Health. 2021 Mar 5;9:526286. doi: 10.3389/fpubh.2021.526286. eCollection 2021. PMID 33748052
- [Derived] Kaar JL, Markovic N, Amsden LB, Gilliland J, Shorter CF, Peters B, Nachreiner NM, Garel M, Nicholas W, Skarpness B, Drews-Botsch C, Hogue CJ, Dabelea D. The Experience of Direct Outreach Recruitment in the National Children's Study. Pediatrics. 2016 Jun;137 Suppl 4(Suppl 4):S258-64. doi: 10.1542/peds.2015-4410G. PMID 27251872
- [Derived] McLaughlin TJ, Aupont O, Kozinetz CA, Hubble D, Moore-Simas TA, Davis D, Park C, Brenner R, Sepavich D, Felice M, Caviness C, Downs T, Selwyn BJ, Forman MR. Multilevel Provider-Based Sampling for Recruitment of Pregnant Women and Mother-Newborn Dyads. Pediatrics. 2016 Jun;137 Suppl 4(Suppl 4):S248-57. doi: 10.1542/peds.2015-4410F. PMID 27251871
- [Derived] Hale DE, Wyatt SB, Buka S, Cherry D, Cislo KK, Dudley DJ, McElfish PA, Norman GS, Reynolds SA, Siega-Riz AM, Wadlinger S, Walker CK, Robbins JM. The National Children's Study: Recruitment Outcomes Using the Provider-Based Recruitment Approach. Pediatrics. 2016 Jun;137 Suppl 4(Suppl 4):S239-47. doi: 10.1542/peds.2015-4410E. PMID 27251870
- [Derived] McGovern PM, Nachreiner NM, Holl JL, Halfon N, Dabelea D, Caulfield L, Cauley JA, Innocenti MS, Amsden L, Markovic N, Riddles M, Adams S. The National Children's Study: Early Recruitment Outcomes Using the Direct Outreach Approach. Pediatrics. 2016 Jun;137 Suppl 4(Suppl 4):S231-8. doi: 10.1542/peds.2015-4410D. PMID 27251869
- [Derived] Trasande L, Andrews HF, Goranson C, Li W, Barrow EC, Vanderbeek SB, McCrary B, Allen SB, Gallagher KD, Rundle A, Quinn J, Brenner B. Early experiences and predictors of recruitment success for the National Children's Study. Pediatrics. 2011 Feb;127(2):261-8. doi: 10.1542/peds.2010-2334. Epub 2011 Jan 24. PMID 21262893